CLINICAL TRIAL: NCT02318498
Title: Stockholm Myocardial Infarction With Normal Coronaries (SMINC)-2
Brief Title: Stockholm Myocardial Infarction With Normal Coronaries (SMINC)-2 Study on Diagnosis Made by Cardiac MRI
Acronym: SMINC-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Medical Research Council (Unknown)
Responsible Party: Principal Investigator, Per Tornvall, Associate professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2
Record Dates: First submitted 2014-12-05; First posted 2014-12-17 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prospective MINCA patients (Active Comparator): Patients with MINCA prospectively investigated with an early CMR with latest technique
  Interventions: Procedure: CMR
- Historical MINCA patients (Placebo Comparator): Patients with MINCA investigated earlier with a late CMR (median 12 days)
  Interventions: Procedure: CMR

INTERVENTIONS:
Procedure: CMR — Intervention performed 2-4 days after admission to hospital with the latest CMR technique including sensitive oedema sequences using T1 mapping

SUMMARY:
Myocardial infarction with angiographically normal coronary arteries (MINCA) is common (7-8 % of all myocardial infarctions). There are several different causes behind MINCA where "true infarction" due to thromboembolism, myocarditis or Takotsubo stress cardiomyopathy are the main findings. The underlying diagnosis is often made by clinical findings sometimes with the help of cardiac MRI (CMR). Investigators have previously shown that it was possible to give 50 % of the patients a diagnosis made by the combination of clinical findings and CMR made in median 12 days after the acute event. The present study aim at improve the diagnostic accuracy by an early CMR with latest technique.

DETAILED DESCRIPTION:
The present study aim at improve the diagnostic accuracy in MINCA with an CMR made 2-4 days after the acute event. The aim is to give 70 % of all patients with MINCA (35-70 years old) a definitive diagnosis made by CMR only. One-hundred and fifty patients will be included and compared with a similar historical sample where 50 % of the patients received a diagnosis made by a late CMR and clinical findings. The study has 80 % power to detect this 20 % absolute difference (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* 35-70 years
* Fullfill the diagnosic criteria of myocardial infarction
* Normal coronary angiography or minor atheromatosis
* Sinus rythm on ECG at admission

Exclusion Criteria:

* Previous myocardial infarction
* Known cardiomyopathy
* Pacemaker or claustrophobia
* Severe chronic obstructive lung or kidney disease
* Pulmonary embolism

Ages: 35 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of an early CMR with the latest technique | 2-4 days after admission
  Show that the more patients get a definite diagnosis (70%) when compared to a historical sample (50%)

SECONDARY OUTCOMES:
Number of patients with correct diagnosis with echocardiography | 12 months
  To study the accuracy of echocardiography compared to CMR using ROC
Number of patients with a postive CT angiography and infarction on CMR | 1 month
  To study CT angiography findings in relation to myocardial infarction shown by CMR
Describe QoL over time | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Per Tornvall, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Steffen Johansson R, Tornvall P, Sorensson P, Nickander J. Reduced stress perfusion in myocardial infarction with nonobstructive coronary arteries. Sci Rep. 2023 Dec 13;13(1):22094. doi: 10.1038/s41598-023-49223-w. PMID 38086910
- [Derived] Sundqvist MG, Sorensson P, Ekenback C, Lundin M, Agewall S, Brolin EB, Cederlund K, Collste O, Daniel M, Jensen J, Y-Hassan S, Henareh L, Hofman-Bang C, Lynga P, Maret E, Sarkar N, Spaak J, Winnberg O, Caidahl K, Ugander M, Tornvall P. CMR Is Often Abnormal Despite Normal Echocardiography in Suspected Myocardial Infarction With Nonobstructed Coronary Arteries. JACC Cardiovasc Imaging. 2023 Dec;16(12):1626-1628. doi: 10.1016/j.jcmg.2023.05.024. Epub 2023 Jul 26. No abstract available. PMID 37498255
- [Derived] Berg E, Agewall S, Brolin EB, Caidahl K, Cederlund K, Collste O, Daniel M, Ekenback C, Jensen J, Y-Hassan S, Henareh L, Maret E, Spaak J, Sorensson P, Tornvall P, Lynga P. Health-related quality-of-life up to one year after myocardial infarction with non-obstructive coronary arteries. Eur Heart J Qual Care Clin Outcomes. 2023 Sep 12;9(6):639-644. doi: 10.1093/ehjqcco/qcac072. PMID 36328780
- [Derived] Sorensson P, Ekenback C, Lundin M, Agewall S, Bacsovics Brolin E, Caidahl K, Cederlund K, Collste O, Daniel M, Jensen J, Y-Hassan S, Henareh L, Hofman-Bang C, Lynga P, Maret E, Sarkar N, Spaak J, Winnberg O, Ugander M, Tornvall P. Early Comprehensive Cardiovascular Magnetic Resonance Imaging in Patients With Myocardial Infarction With Nonobstructive Coronary Arteries. JACC Cardiovasc Imaging. 2021 Sep;14(9):1774-1783. doi: 10.1016/j.jcmg.2021.02.021. Epub 2021 Apr 14. PMID 33865778
- [Derived] Tornvall P, Brolin EB, Caidahl K, Cederlund K, Collste O, Daniel M, Ekenback C, Jensen J, Y-Hassan S, Henareh L, Hofman-Bang C, Lynga P, Maret E, Sarkar N, Spaak J, Sundqvist M, Sorensson P, Ugander M, Agewall S. The value of a new cardiac magnetic resonance imaging protocol in Myocardial Infarction with Non-obstructive Coronary Arteries (MINOCA) - a case-control study using historical controls from a previous study with similar inclusion criteria. BMC Cardiovasc Disord. 2017 Jul 24;17(1):199. doi: 10.1186/s12872-017-0611-5. PMID 28738781